CLINICAL TRIAL: NCT01298219
Title: A Multicenter, Randomized, Placebo-controlled, Double-blinded Study of the Efficacy and Safety of Lubiprostone in Subjects With Opioid-induced Bowel Dysfunction
Brief Title: Opioid-induced Bowel Dysfunction (OBD) Pivotal Assessment of Lubiprostone (OPAL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Sucampo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OBD1033
Record Dates: First submitted 2011-01-20; First posted 2011-02-17 (Estimated); Results first posted 2019-12-24 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2013-02

CONDITIONS: Opioid-induced Bowel Dysfunction
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Care provider and outcomes assessor were also blinded for this double-blind trial.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone (Experimental): 24 mcg capsules twice daily (BID)
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator): 0 mcg capsules twice daily (BID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — 24 mcg administered orally twice daily (BID)
  Other Names: Amitiza
  Arms: Lubiprostone
Drug: Placebo — Matching placebo, 0 mcg administered orally twice daily (BID)
  Other Names: No other names
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to evaluate the efficacy and safety of lubiprostone administration in subjects with Opioid-induced Bowel Dysfunction.

ELIGIBILITY:
Inclusion Criteria:

A patient can be considered for eligibility to participate if he/she:

* Has been consistently treated for chronic, noncancer-related pain with any oral, transdermal, intravenous, or subcutaneous opioid for at least 30 days prior to screening
* Is diagnosed with OBD
* Is capable of utilizing an electronic diary to report daily spontaneous bowel movements (SBMs)
* Is willing to continue opioid therapy and discontinue the use of laxatives, stool softeners, and other concomitant medications affecting gastrointestinal motility throughout the study

Exclusion Criteria:

A patient cannot be considered for eligibility to participate if he/she:

* Uses opioids for the treatment of cancer-related pain, abdominal pain, mechanical bowel obstructions, bowel disorders, and constipation not arising from opioid use, but instead attributable to dietary, neurologic, congenital, or endocrine disorders, scleroderma, and/or for the management of drug addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Mallinckrodt
Locations (141):
- United States (114):
  - North Alabama Research Center, Athens, Alabama
  - Innovative Clinical Trials, Inc., Birmingham, Alabama
  - Achieve Clinical Research, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - G&L Research, LLC, Foley, Alabama
  - Healthscan Research, Montgomery, Alabama
  - River Region Research, Tallassee, Alabama
  - Anasazi Internal Medicine PC, Phoenix, Arizona
  - Aureas Research, Inc, Little Rock, Arkansas
  - Certified Clinical Research, Carmichael, California
  - California Clinical Research, Inc., Davis, California
  - Family Medical Center, Foothill Ranch, California
  - South Orange County Surgical Medical Group, Laguna Hills, California
  - Clinical Trials Research, Lincoln, California
  - Clear Vision Research, Long Beach, California
  - Long Beach VA Medical Center, Long Beach, California
  - Clear Vision Research, Los Angeles, California
  - Facey Medical Foundation, Mission Hills, California
  - North County Clinical Research, Oceanside, California
  - SDS Clinical Trials, Inc., Orange, California
  - Probe Clinical Research Corporation, Riverside, California
  - Probe Clinical Research Corporation - Santa Ana, Santa Ana, California
  - Westlake Medical Research, Westlake Village, California
  - Mountain View Clinical Research, Denver, Colorado
  - Meridien Research, Bradenton, Florida
  - Coastal Orthopedics & Pain Management, Bradenton, Florida
  - Florida Research & Testing, LLC, Clearwater, Florida
  - Avail Clinical Research, DeLand, Florida
  - S&W Clinical Research, Fort Lauderdale, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Physicians Regional Medical Group, Naples, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Paddock Park Clinical Research, Ocala, Florida
  - Journey Research, Inc., Oldsmar, Florida
  - Compass Research, Orlando, Florida
  - Andres Patron, DO, PA, Pembroke Pines, Florida
  - Advent Clinical Research Centers, Pinellas Park, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - Orthopedic Research Institite, Royal Palm Beach, Florida
  - IC Research, Sanford, Florida
  - Sarasota Memorial Pain Care Center, Sarasota, Florida
  - Tampa Clinical Research, Tampa, Florida
  - Southeastern Regional Research Group, Columbus, Georgia
  - Better Health Clinical Research, Newnan, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Sonora Clinical Research, Boise, Idaho
  - Nautical Clinical Research, Meridian, Idaho
  - Anesthesia/Pain Control Indiana University School of Medicine, Chicago, Illinois
  - Knight Center for Integrated Health, Peoria, Illinois
  - Ridge Family Practice, Council Bluffs, Iowa
  - Lee Research Institute, Lenexa, Kansas
  - Kentucky Medical Research Center, Lexington, Kentucky
  - Bluegrass Internal Medicine, Owensboro, Kentucky
  - Horizon Research Group, Baton Rouge, Louisiana
  - Miray Medical Center, Brockton, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Coastal Research, Weymouth, Massachusetts
  - Ashok Jain, MD, Dearborn, Michigan
  - Shores Medical Associates, Saint Clair Shores, Michigan
  - Mid-America Clinical Research LLC, St Louis, Missouri
  - Montana Medical Research, Inc., Missoula, Montana
  - Independent Clinical Researchers, Las Vegas, Nevada
  - AB Clinical Trials, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Clinical Research Advantage, Inc., Las Vegas, Nevada
  - Lab2Marche, Las Vegas, Nevada
  - Aloha Medical Center, Las Vegas, Nevada
  - Edison Medical Group, Edison, New Jersey
  - Clinical Research Program, Marlton, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Drug Trials America, Hartsdale, New York
  - Family Health Medical Services PLLC, Jamestown, New York
  - U of Rochester, Rochester, New York
  - Medical Frontiers, Carlisle, Ohio
  - Hightop Medical Research Center, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Parsons Avenue Medical Center, Columbus, Ohio
  - Hometown Urgent Care, Groveport, Ohio
  - Northstar Medical Research, LLC, Middleburg Heights, Ohio
  - Pharmacotherpy Research Associates Inc, Zanesville, Ohio
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Sunstone Medical Research, Medford, Oregon
  - Fanno Creek Clinic, Portland, Oregon
  - McMillen & Magargle, Mechanicsburg, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Hartwell Research Group, Anderson, South Carolina
  - Degarmo Institute of Medical Research, Greer, South Carolina
  - Pain Specialists of Charleston, North Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - InvestiClin Research, Brentwood, Tennessee
  - SCRI Research Center, Germantown, Tennessee
  - Prevention & Strengthening Solutions, Inc., Humboldt, Tennessee
  - FutureSearch Trials of Neurology & Sleep Lab, Austin, Texas
  - Jaron Winston, MD, Austin, Texas
  - KRK Medical Research, Dallas, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Pillar Clinical Research, LLC, Dallas, Texas
  - Galenos Research, Dallas, Texas
  - Diversified Medical Practice, P.A., Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Dependable Clinical Research, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Bobby Huynh, Richardson, Texas
  - Sun Research Institute, San Antonio, Texas
  - Spring Clinical Research, Sugar Land, Texas
  - Pioneer Research Solutions, Sugar Land, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - ACR Research Salt Lake City, West Jordan, Utah
  - Virginia Research Center, LLC, Midlothian, Virginia
- Belgium (3):
  - Pain Clinic-Heilig Hart Ziekenhuis Roeselare, Roeselare, Westlaan 123
  - Huisartsenpraktijk De Regenboog, Antwerp
  - Dr Capiau - GP Practice, Wetteren
- Czechia (7):
  - St. Anne's University Hospital - centrum pro, Brno
  - Nemocnice Jablonec nad Nisou, p.o., Jablonec nad Nisou
  - Ambulance bolesti, Krajska nemocnice Liberec, Liberec
  - Klaudianova nemocnice Mlada Boleslav, Mladá Boleslav
  - Clintrial s.r.o., Prague
  - Neurologicka ambulance, Prague
  - Regional Hospital T. B., a.s., Zlín
- Germany (3):
  - Schmerzzentrum Berlin, Berlin
  - Schmerztherapeutische- Ärztezentrum Nordstadt, Hanover
  - Schmerz und Palliativzentrum, Wiesbaden
- NZOZ Dom Sue Ryder prowadzony przez Pallmed Sp. z o.o., Bydgoszcz, Poland
- Sweden (3):
  - Hagakliniken, Gothenburg
  - Karolinska University Hospita- Dept of Anaesthesia, Pain Div., Stockholm
  - S3 Clinical Research Centers, Vällingby
- United Kingdom (10):
  - ElyBridge Surgery, Ely, Cardiff
  - Randalstown Medical Practice, Randalstown, Co Antrim
  - Sea Road Surgery, Bexhill-on-Sea, E.Sussex
  - Sheepcot Medical Centre,, Watford, Herts
  - Fylde Coast Clinical Research Ltd, Blackpool, Lancsashire
  - Ballygomartin Group Practice, Belfast, Northern Ireland
  - The Waterfront Medical Centre, Barry, Wales
  - Valleyfield Health Center, Dunfermline
  - Frome Medical Practice, Frome
  - Mortimer Surgery, Reading

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 07 December 2010 to 16 November 2011 Recruitment sites: 91 U.S. investigative sites and 14 E.U. investigative sites
Pre-assignment Details: Safety evaluable population includes all subjects who were randomized and dosed. Intention to treat (ITT) population includes only those subjects who were dosed and provided at least one post-treatment efficacy assessment.
Period: Overall Study
Arm/Group | Lubiprostone | Placebo
Started | 219 | 220
Intention to Treat (ITT) | 219 | 220
Safety Analysis Set | 219 | 220
Completed | 169 | 184
Not Completed | 50 | 36

BASELINE CHARACTERISTICS:
Population: Baseline analysis based on ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubiprostone | Placebo | Total
Number analyzed (Participants) | 219 | 220 | 439
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (9.01) | 51.5 (11.68) | 51.7 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 138 | 276
  Male | 81 | 82 | 163
Region of Enrollment [Number; unit: participants]
  Czech Republic | 6 | 8 | 14
  Belgium | 2 | 2 | 4
  United States | 202 | 203 | 405
  Poland | 2 | 2 | 4
  United Kingdom | 3 | 2 | 5
  Germany | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified as Treatment Responders Within 12 Weeks
Description: Spontaneous bowel movement (SBM) is defined as any BM that does not occur within 24 hours after use of rescue medication. To be classified as responders, participants are required to demonstrate at least moderate response (≥ 1 SBM improvement over baseline SBM frequency) for all treatment weeks for which observed data are available, and must additionally demonstrate a full response (≥ 3 SBMs per week) for at least 9 of the 12 treatment weeks.
Time Frame: 12 weeks
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 219 | 220
Participants | 59 | 41

2. Secondary Outcome: Number of SBMs Per Week at Week 8
Time Frame: at Week 8
Population: Intention to treat with data at Week 8
Measure: Mean (Standard Deviation); unit: SBMs/week
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 168 | 182
SBMs/week | 2.9 (3.18) | 2.5 (3.03)

3. Secondary Outcome: Number of Participants Who Experienced First SBM Within 48 Hours After Dose Initiation
Time Frame: within 48 hours post-dose
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 219 | 220
Participants
  within 24 Hours | 110 | 84
  within 48 Hours | 157 | 134

4. Secondary Outcome: Number of SBMs Per Week at Week 12
Time Frame: at Week 12
Population: Intention to treat with data at Week 12
Measure: Mean (Standard Deviation); unit: SBMs/week
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 159 | 180
SBMs/week | 3.1 (3.13) | 2.7 (3.34)

5. Secondary Outcome: Number of SBMs Per Week Overall
Description: Overall is defined as the length of time from first dose to last follow-up within 2 weeks after last dose.
Time Frame: within 14 weeks
Population: Intention to treat with data at Week 14
Measure: Mean (Standard Deviation); unit: SBMs/week
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 213 | 218
SBMs/week | 4.3 (2.96) | 3.7 (2.53)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs): 14 weeks (from time of first dose to 14 days post-treatment)
Description: Number of participants at risk represents the Safety Evaluable population. Safety Evaluable population includes all subjects who were randomized and dosed. ITT population (in Participant Flow) includes only subjects who dosed and provided at least one post-treatment efficacy assessment.
Arm/Group | Lubiprostone | Placebo
All-Cause Mortality (participants affected / at risk) | 1/219 | 0/220
Serious Adverse Events (participants affected / at risk) | 7/219 | 6/220
Other Adverse Events (participants affected / at risk) | 72/219 | 44/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lubiprostone (N=219) | Placebo (N=220)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Fecaloma (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Drug Toxicity (Injury, poisoning and procedural complications) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lubiprostone (N=219) | Placebo (N=220)
Diarrhea (Gastrointestinal disorders) | 24 | 8
Nausea (Gastrointestinal disorders) | 21 | 10
Vomiting (Gastrointestinal disorders) | 9 | 11
Abdominal Pain (Gastrointestinal disorders) | 15 | 0
Flatulence (Gastrointestinal disorders) | 6 | 5
Urinary Tract Infection (Infections and infestations) | 7 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Gamma-Glutamyltransferase Increased (Investigations) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No